CLINICAL TRIAL: NCT05177510
Title: Mifepristone Outpatient Labour Induction
Acronym: MOLI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CW003; 2021-004860-93 (EudraCT Number)
Record Dates: First submitted 2021-11-17; First posted 2022-01-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Labor, Induced
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Intervention Model Description: Double-blinded parallel group randomised control trial. Intervention arm Mifepristone plus standard care, comparator arm placebo plus standard of care .
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double parallel group randomised control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mifepristone and standard of care (Experimental): Mifepristone 300mg once only and standard of care
  Interventions: Drug: Mifepristone
- Placebo (Placebo Comparator): Placebo 300mg once only and standard of care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mifepristone — Progestin Antagonist
  Arms: Mifepristone and standard of care
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The number of women having an induction of labour is increasing and is currently used in 33% of pregnancies for a range of medical reasons. The majority of women are admitted to hospital to have their labour induced, using methods which are protracted and associated with a poor birth experience, making them both costly and unpopular. Further, current methods of outpatient induction are unsuitable, unsafe and/or have a poor acceptability. The COVID-19 pandemic has driven a reduction in the number of face-to-face interactions taking place across all areas of medicine. Proving the efficacy and safety of Mifepristone would significantly reduce pre-labour admission rates and hospital length of stay for pregnant women, who are at particularly higher risk of COVID-19, and reduce delivery costs.

DETAILED DESCRIPTION:
The study is a double blinded, two arms, multi-centre randomised controlled clinical trial to investigate the clinical effectiveness, safety and resource utilisation of intervention for the induction of labour in women admitted to the hospital. Subjects will be randomised 1:1 to one of the two arms to receive:

Arm 1: Mifepristone + standard of care Arm 2: Placebo + standard of care

The study treatment will commence from the administration of the Mifepristone or placebo. The participants will be assessed 2 days after treatment regimen will be completed as an in-patient.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 36+5 and 41+5 weeks of gestation
2. Singleton pregnancy
3. Aged 18 years or older
4. Unfavourable cervix (Bishop Score less than or equal to 6)
5. The ability to understand and sign a written informed consent form, prior to participation in any screening procedures and must be willing to comply with all study requirements.

Exclusion Criteria:

1. Breech presentation
2. Early labour
3. Contraindication to vaginal birth (placenta praevia, transverse lie, known or suspected cephalo-pelvic disproportion or other factor contraindicated to vaginal birth in the opinion of the investigator)
4. Fetal growth restriction with oligohydramnios and/or abnormal Dopplers
5. Presence of reduced fetal movements requiring urgent delivery, abnormal CTG or recent antepartum haemorrhage requiring immediate delivery
6. Medical conditions:

   i. sexually transmitted infections (active infections only) ii. bleeding disorders, on anticoagulants, steroid or aspirin therapy iii. prior uterine operations (Caesarean Section or myomectomy)
7. Contra-indications to mifepristone including chronic adrenal, hepatic, renal failure
8. Hypersensitivity to mifepristone or to any excipients, or malnutrition
9. Severe asthma uncontrolled by therapy and inherited porphyria
10. Any investigational drug with an expected interaction with mifepristone which has been administered within 30 days prior to the trial drug administration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women between 36+5 and 41+5 weeks of gestation.
Enrollment: 400 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure of women in labour or delivered within 2 days of intervention | up to 2 days after administration of intervention
  To determine proportion of women who do not require an induction of labour within 2 days of intervention with mifepristone (superiority).

SECONDARY OUTCOMES:
Change in clinical outcomes | up to 6 weeks after delivery
  Occurrence of changes in clinical outcomes such as cervical ripening and interval to delivery.
Determine whether intervention reduces resource utilisation and patient experience | after delivery and up to 6 weeks after delivery
  Patient reported outcomes will be collected following administration of questionnaires after delivery and up to 6 weeks after delivery
To assess the efficacy and safety of Mifepristone for the outpatient induction of labour | up to 6 weeks after delivery
  Incidence and severity of adverse events in maternal and neonatal

CONTACTS AND LOCATIONS:
Overall Officials: Mark Johnson, Study Chair — Chelsea and Westminster NHS Foundation Trust; Damon Foster, Study Director — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Research team wishes to enable any meta-analyses of such trials making appropriate requests. No plan to share IPD has been made at this time.